CLINICAL TRIAL: NCT05931783
Title: Randomized Comparison of HARVesting the Left Internal Thoracic Artery in a Skeletonized Versus Pedicled Technique: the HARVITA Trial
Brief Title: Randomized Comparison of Skeletonized Versus Pedicled Left Internal Thoracic Artery
Acronym: HARVITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1135/2023
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease
Keywords: CABG; LITA; graft patency; skeletonized vs. pedicled
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skeletonized harvesting technique (Active Comparator): In skeletonized harvesting technique, only the left internal artery itself is harvested.
  Interventions: Procedure: skeletonized harvesting technique
- pedicled harvesting technique (Active Comparator): In pedicled harvesting technique the left internal thoracic artery, it's accompanying veins and parts of the endothoracic fascia is harvested, creating a 1-2 cm broad pedicle.
  Interventions: Procedure: pedicled harvesting technique

INTERVENTIONS:
Procedure: skeletonized harvesting technique — In patients who are randomized to this treatment arm, the left internal thoracic artery will be harvested in skeletonized technique. Thereby, only the artery itself is harvested.
  Arms: skeletonized harvesting technique
Procedure: pedicled harvesting technique — In patients who are randomized to this treatment arm, the left internal thoracic artery will be harvested in pedicled technique. Thereby, the artery will be harvested together with the accompanying veins, the endothoracic fascia and fatty tissue in order to create an 1-2 cm broad pedicle.
  Arms: pedicled harvesting technique

SUMMARY:
Internal thoracic arteries can be harvested in skeletonized or pedicled technique. Latest research has posed a potential adverse effect of skeletonizing the internal thoracic arteries on graft patency rates and clinical outcome. Prospective, randomized, multi-centre trials are necessary to investigate the impact of harvesting technique of left internal thoracic artery (LITA) on graft patency rates and clinical outcome after coronary artery bypass grafting.

The HARVITA trial compares skeletonized and pedicled harvesting technique of LITA regarding graft patency rates and patient survival.

ELIGIBILITY:
Inclusion criteria:

Primary isolated CABG patients with multi-vessel disease (defined as ≥70 % stenosis of the left anterior descending artery (LAD) and ≥50% stenosis of circumflex and right coronary territory, with or without a ≥50% stenosis of the left main artery).

Exclusion criteria:

* Age > 80 years
* Planned CABG without LITA use
* Preoperative mediastinal radiation therapy
* Emergency operation
* Minimal invasive coronary artery bypass surgery
* Any concomitant cardiac or non-cardiac procedures
* Previous cardiac surgery
* Known contrast agent allergy
* Severe stenosis of the left subclavian artery/ left-sided subclavian steal syndrome
* Chronic kidney disease (GFR <60ml/min/1.73m²)
* Life expectancy of less than 5 years
* Pregnancy
* Hyperthyroidism
* Iodine allergy

Intraoperative exclusion criteria:

* Y/T graft off the LITA graft
* LITA sequential grafting
* LITA target vessel other than LAD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Death or LITA graft occlusion in cCTA or invasive angiography within 2 years (+/- 3 months) after surgery. | 2 years (+/- 3 months) after surgery
  The primary endpoint will be compared between the two treatment groups using Kaplan-Meier graphs and a center stratified two sample log-rank test. In addition, Cox proportional hazards regression analysis adjusting for clinically relevant confounders will be performed. Hazard ratios and their 95% confidence intervals will be estimated.
  LITA graft occlusion is defined as the absence of contrast detection in the lumen of the graft indicating a 100% occlusion of LITA graft.

SECONDARY OUTCOMES:
composite outcome of all-cause death, myocardial infarction and repeated revascularization | 1 year, 2 years and 5 years after surgery
  The composite outcome of all-cause death, myocardial infarction and repeated revascularization will be compared with Kaplan-Meier graphs together with log-rank testing.

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Abfalterer, Dr. med. univ., Principal Investigator — Medical University Innsbruck; Nikolaos Bonaros, Univ. Prof. Dr., Principal Investigator — Medical University Innsbruck
Locations (8):
- Austria (3):
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Germany (4):
  - University of Duisburg-Essen, Essen
  - University of Freiburg, Freiburg im Breisgau
  - University Hospital Gießen, Giessen
  - University of Jena, Jena
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] Lamy A, Browne A, Sheth T, Zheng Z, Dagenais F, Noiseux N, Chen X, Bakaeen FG, Brtko M, Stevens LM, Alboom M, Lee SF, Copland I, Salim Y, Eikelboom J; COMPASS Investigators. Skeletonized vs Pedicled Internal Mammary Artery Graft Harvesting in Coronary Artery Bypass Surgery: A Post Hoc Analysis From the COMPASS Trial. JAMA Cardiol. 2021 Sep 1;6(9):1042-1049. doi: 10.1001/jamacardio.2021.1686. PMID 34132753
- [Background] Gaudino M, Audisio K, Rahouma M, Chadow D, Cancelli G, Soletti GJ, Gray A, Lees B, Gerry S, Benedetto U, Flather M, Taggart DP; ART Investigators. Comparison of Long-term Clinical Outcomes of Skeletonized vs Pedicled Internal Thoracic Artery Harvesting Techniques in the Arterial Revascularization Trial. JAMA Cardiol. 2021 Dec 1;6(12):1380-1386. doi: 10.1001/jamacardio.2021.3866. PMID 34586338